CLINICAL TRIAL: NCT00781274
Title: A Phase 3 Study of MP-424 in Combination With Peginterferon Alfa-2b and Ribavirin (RBV) in Subjects With (Genotype 1) Hepatitis C Who Did Not Respond to Previous Treatment
Brief Title: Efficacy and Safety of MP-424, Peginterferon Alfa-2b and Ribavirin in Chronic Hepatitis C Who Have Not Achieved an Undetectable HCV RNA Level With Previous Interferon Based Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G060-A9
Record Dates: First submitted 2008-10-24; First posted 2008-10-28 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Ribavirin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MP-424 (Experimental)
  Interventions: Drug: MP-424; Drug: Ribavirin; Drug: Peginterferon Alfa-2b

INTERVENTIONS:
Drug: MP-424 — 750 mg every 8 hours for 12 weeks
  Other Names: Telaprevir
Drug: Ribavirin — 600 - 1000 mg/day based on body weight for 24 weeks
Drug: Peginterferon Alfa-2b — 1.5 mcg/kg/week for 24 weeks

SUMMARY:
This study will evaluate the efficacy and safety of MP-424 with Peginterferon Alfa-2b and RBV in patients with (Genotype 1) hepatitis C, who did not respond to previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 1, chronic hepatitis C
* Non-responders (patient who did not respond to previous treatment)
* Able and willing to follow contraception requirements

Exclusion Criteria:

* Cirrhosis of the liver or hepatic failure
* Hepatitis B surface antigen-positive or HIV antibodies-positive
* History of, or concurrent hepatocellular carcinoma
* History of, or concurrent depression, schizophrenia; or suicide attempt in the past
* Pregnant, lactating, or suspected pregnant patients, or male patients whose female partner is pregnant

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fumitaka Suzuki, MD, Principal Investigator — Department of Hepatology, Toranomon Hospital
Locations (1):
- Toranomon Hospital, Kawasaki, Takatsu-ku, Japan

REFERENCES:
- [Result] Hayashi N, Okanoue T, Tsubouchi H, Toyota J, Chayama K, Kumada H. Efficacy and safety of telaprevir, a new protease inhibitor, for difficult-to-treat patients with genotype 1 chronic hepatitis C. J Viral Hepat. 2012 Feb;19(2):e134-42. doi: 10.1111/j.1365-2893.2011.01528.x. Epub 2011 Nov 8. PMID 22239511

RESULTS

PARTICIPANT FLOW:
Groups:
- MP-424: Drug: MP-424 750 mg every 8 hours for 12 weeks Other Name: Telaprevir
  Drug: Ribavirin 600 - 1000 mg/day based on body weight for 24 weeks
  Drug: Peginterferon Alfa-2b 1.5 mcg/kg/week for 24 weeks
Period: Overall Study
Arm/Group | MP-424
Started | 32
Completed | 30
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | MP-424
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Achieving Undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at 24 Weeks After Completion of Drug Administration (SVR, Sustained Viral Response)
Time Frame: After 24 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving SVR
Arm/Group | MP-424
Number analyzed (Participants) | 32
percentage of subjects achieving SVR | 34.4 [18.6 to 53.2]

ADVERSE EVENTS:
Arm/Group | MP-424
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-424 (N=32)
Vomiting (Gastrointestinal disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Malaise (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP-424 (N=32)
Nasopharyngitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Anaemia (Blood and lymphatic system disorders) | 32
Hyperthyroidism (Endocrine disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 15
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 11
Headache (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 6
Dry eye (Eye disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 3
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 16
Alopecia (Skin and subcutaneous tissue disorders) | 7
Drug eruption (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Rash papular (Skin and subcutaneous tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pyrexia (General disorders) | 30
Malaise (General disorders) | 22
Injection site erythema (General disorders) | 2
Injection site reaction (General disorders) | 3
Influenza like illness (General disorders) | 2
Thirst (General disorders) | 2
Injection site pruritus (General disorders) | 3
White blood cell count decreased (Investigations) | 22
Platelet count decreased (Investigations) | 22
Blood uric acid increased (Investigations) | 25
Hyaluronic acid increased (Investigations) | 15
Blood creatinine increased (Investigations) | 12
Blood bilirubin increased (Investigations) | 10
Blood triglycerides increased (Investigations) | 8
Blood phosphorus decreased (Investigations) | 6
Blood potassium decreased (Investigations) | 3
Laboratory test abnormal (Investigations) | 3
Protein urine present (Investigations) | 2
Low density lipoprotein increased (Investigations) | 2
Blood thyroid stimulating hormone increased (Investigations) | 2
Blood calcium decreased (Investigations) | 2
Lipids abnormal (Investigations) | 2
Transaminases increased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other